CLINICAL TRIAL: NCT02208089
Title: A Prospective Trial of Simultaneous Combined Transepithelial Photorefractive Keratectomy and Corneal Collagen Cross-linking for Keratoconus
Brief Title: Simultaneous TransPRK and Corneal Collagen Cross-Linking
Acronym: TransPRKCXL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bruce Allan (Other)
Collaborators: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor-Investigator, Bruce Allan, Consultant Ophthalmic Surgeon, Moorfields Eye Hospital NHS Foundation Trust
Organization: Moorfields Eye Hospital NHS Foundation Trust (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ALLB1018
Record Dates: First submitted 2014-07-25; First posted 2014-08-04 (Estimated); Results first posted 2019-02-08 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2018-09

CONDITIONS: Keratoconus
Keywords: Keratoconus; Corneal collagen cross-linking; Photorefractive keratectomy
MeSH Terms: conditions — Keratoconus | interventions — Corneal Cross-Linking

STUDY DESIGN:
Intervention Model Description: Interventional case series with matched historical controls
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TransPRKCXL (Experimental): Simultaneous combined transepithelial photorefractive keratectomy (TransPRK) and corneal collagen cross-linking (CXL)
  Interventions: Procedure: Transepithelial Photorefractive Keratectomy (TransPRK); Procedure: Corneal Collagen Cross-Linking (CXL)
- CXL only (Active Comparator): Corneal collagen cross-linking (CXL) using the same protocol without transepithelial photorefractive keratectomy
  Interventions: Procedure: Corneal Collagen Cross-Linking (CXL)

INTERVENTIONS:
Procedure: Transepithelial Photorefractive Keratectomy (TransPRK) — Aberrometry or topography guided transepithelial photorefractive keratectomy (TransPRK) using the Schwind Amaris 750s excimer laser (www.eye-tech-solutions.com), an 8mm treatment diameter, and a tissue saving algorithm targeting selected higher order aberrations only. TransPRK will be followed immediately by corneal collagen cross-linking (CXL).
  Other Names: Corneal surface excimer laser treatment
  Arms: TransPRKCXL
Procedure: Corneal Collagen Cross-Linking (CXL) — Riboflavin soak: 10 minutes total soak time; application of 0.1% riboflavin preparation (VibeX Rapid - www.avedro.com) each 2 minutes with gentle balanced salt solution irrigation to remove excess riboflavin prior to UV light exposure.
  UV light exposure: Total treatment time 8 minutes (370nm wavelength; 30mW/cm2 irradiance; 4 minutes total UV exposure time, pulsed 1.5 seconds on 1.5 seconds off; Avedro KXL I light source)
  Other Names: Rapid corneal collagen cross-linking

SUMMARY:
Young patients with keratoconus face two problems: disease progression and corneal shape irregularity leading to poor vision even in spectacles.

Corneal collagen cross-linking (CXL) is a new treatment designed to halt disease progression in keratoconus. The aim is to stiffen the cornea thereby preventing further shape deterioration.

Topography or wavefront guided transepithelial photorefractive keratectomy (transPRK) uses the excimer laser (the laser used to correct sight in 'laser eye surgery') to reduce corneal shape irregularity in early stage keratoconus, reducing dependence on contact lenses.

In transPRK, the corneal skin layer is removed in a well controlled, no touch procedure, preparing the cornea for CXL. Performing both treatments simultaneously (combining both procedures in one operation) may offer several advantages over performing CXL first then waiting for corneal shape to stabilise before performing transPRK. In particular, visual rehabilitation may be faster. This study aims to evaluate visual recovery after simultaneous CXL and transPRK in progressive early stage keratoconus. Visual recovery in these patients will be compared with results for a similar group of patients with early stage keratoconus who have already been treated with CXL alone.

DETAILED DESCRIPTION:
Features which distinguish this trial from previous trials of combined photorefractive keratectomy (PRK) and corneal collagen cross-linking (CXL) are: a rapid, pulsed light, CXL protocol; and a treatment programming algorithm for PRK designed to target higher order aberrations only with no compensatory additional laser corneal tissue removal.

Excimer laser treatment will be performed with the Schwind Amaris 750S laser (www.eye-tech-solutions.com). Unique features of this system utilised here include:

* Pre-programmed transepithelial ablation - laser removal of the minimum area of corneal epithelium required for PRK promoting more rapid recovery than conventional methods (20% alcohol application and manual epithelial removal). An 8mm diameter ablation zone will be applied throughout.
* Enhanced algorithms for minimal laser tissue removal - in this trial, the investigators are targeting higher order aberrations only (coma in particular) with the aim of improving spectacle corrected visual acuity without regard to the predicted spherocylindrical outcome. Unlike other current excimer laser platforms, Schwind Amaris treatment programming software allows treatment for irregular astigmatism without additional compensatory laser tissue removal to correct the spherocylindrical change induced by treatment of higher order aberrations. Higher order aberrations can also be treated selectively. The investigators will use an algorithm step that targets only aberrations (up to 6th order Zernike polynomials) with a value greater than 2 standard deviations from the population mean in normative data. These treatment planning steps allow the laser to create a large diameter treatment with minimal treatment depth.

Laser epithelial removal alone (transPTK at depth 55µm) removes a maximum 65µm of tissue in the corneal periphery. For patients with 390µm at the thinnest point, transPTK will therefore leave above 325µm residual stromal thickness prior to CXL. This is in line with recommendations for minimum stromal thickness after epithelial removal in the CXL protocol used here. Limited stromal reshaping is achieved in this simple embodiment of transPRK for keratoconus by taking advantage of the masking effect of the corneal epithelium, which tends to be thinnest over the cone apex. Where the thinnest point is greater than 390µm, further reductions in corneal shape irregularity can be produced by adding either wavefront or topography guided additional stromal ablation using custom programming on the Schwind Amaris laser. Ocular wavefront (aberrometry) guided smoothing will be used for patients with a 5.5mm or larger pupil at scanning and a consistent scan sequence (3 scans within 0.5 dioptre (D) spherical equivalent refraction). Corneal wavefront (topography) guided smoothing will be used for patients with ocular wavefront scans which do not meet these criteria. In all cases, a minimum corneal stromal thickness prior to CXL of 325µm will be preserved.

Immediately after PRK, corneal collagen cross-linking will be performed using the following protocol

Riboflavin soak: 10 minutes total soak time; application of 0.1% riboflavin preparation (VibeX Rapid - www.avedro.com) each 2 minutes with gentle balanced salt solution irrigation to remove excess riboflavin prior to UV light exposure.

UV light exposure: Total treatment time 8 minutes (370nm wavelength; 30mW/cm2 irradiance; 4 minutes total UV exposure time, pulsed 1.5 seconds on 1.5 seconds off; Avedro KXL I light source)

Mitomycin C will not be used. A bandage contact lens will be applied at the end of treatment and a standard post photorefractive keratectomy topical and systemic drug treatment regimen will be used in every case with initial clinical review 1 week after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with progressive stage II or III keratoconus
* CDVA < 0.00 logMAR or subjective problems with spectacle corrected visual quality (ghost images or light scatter symptoms)

Exclusion Criteria:

* Active ocular surface disease
* Minimum corneal thickness <390µm (leaving 325µm residual stromal thickness after transPTK - in line with minimum thickness recommendations for the study CXL protocol)
* Vulnerable groups (patients whose capacity for giving informed consent to participate in the trial may be impaired)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2014-08; Primary Completion 2016-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce D Allan, MD FRCOphth, Principal Investigator — Moorfields Eye Hospital NHS Foundation Trust; Dan M Gore, FRCOphth, Principal Investigator — Moorfields Eye Hospital NHS Foundation Trust
Locations (1):
- Moorfields Eye Hospital NHS Foundation Trust, 162 City Road, London, United Kingdom

REFERENCES:
- [Background] Gore DM, Shortt AJ, Allan BD. New clinical pathways for keratoconus. Eye (Lond). 2013 Mar;27(3):329-39. doi: 10.1038/eye.2012.257. Epub 2012 Dec 21. PMID 23258309
- [Background] Kanellopoulos AJ, Asimellis G. Keratoconus management: long-term stability of topography-guided normalization combined with high-fluence CXL stabilization (the Athens Protocol). J Refract Surg. 2014 Feb;30(2):88-93. doi: 10.3928/1081597X-20140120-03. PMID 24763473

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with Stage I-III keratoconus and corrected vision <20/20 were recruited. Recruitment period: August 2014-July2015. Location: dedicated keratoconus clinic at Moorfields Eye Hospital, London.
Pre-assignment Details: 63 eligible patients were screened; 11 declined to participate after discussing consent information; 5 patients were found to be ineligible because of insufficient residual corneal stromal depth following PRK programming, leaving 47 patients who were treated with TransPRK/CXL
Groups:
- TransPRKCXL: Simultaneous combined transepithelial photorefractive keratectomy (TransPRK) and corneal collagen cross-linking (CXL)
  Transepithelial Photorefractive Keratectomy (TransPRK): Aberrometry or topography guided transepithelial photorefractive keratectomy (TransPRK) using the Schwind Amaris 750s excimer laser (www.eye-tech-solutions.com), an 8mm treatment diameter, and a tissue saving algorithm targeting selected higher order aberrations only. TransPRK will be followed immediately by corneal collagen cross-linking (CXL).
  Corneal Collagen Cross-Linking (CXL): Riboflavin soak: 10 minutes total soak time; application of 0.1% riboflavin preparation (VibeX Rapid - www.avedro.com) each 2 minutes with gentle balanced salt solution irrigation to remove excess riboflavin prior to UV light exposure.
  UV light exposure: Total treatment time 8 minutes (370nm wavelength; 30mW/cm2 irradiance; 4 minutes total UV exposure time, pulsed 1.5 seconds on 1.5 seconds off; Avedro KXL I light source)
- CXL Only: Patients treated with standard accelerated corneal collagen cross-linking (historical controls)
Period: Overall Study
Arm/Group | TransPRKCXL | CXL Only
Started | 47 | 47
Completed | 40 | 47
Not Completed | 7 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 6 | 0

BASELINE CHARACTERISTICS:
Population: Matched historical control cases of CXL treated using the same CXL protocol as the TransPRKCXL group prior to commencement of recruitment. These control cases were consecutive cases with 2 year follow up data, matched for age, corneal pachymetry, and corneal curvature with the TransPRK group
Groups:
- CXL Only: Corneal collagen cross-linking (CXL), manual corneal epithelial removal, no excimer laser treatment
  CXL protocol was identical in both study arms. After corneal epithelial removal, a 10 minute soak with Vibex rapid (www.avedro.com) was followed by 8 minutes pulsed UV light using a uniform beam source (KXL - www.avedro.com) and a 1.5 second on/off cycle (7.2mJ/cm2 total energy @ 30mW/cm2 irradiance).
- Total: Total of all reporting groups
Arm/Group | TransPRKCXL | CXL Only | Total
Number analyzed (Participants) | 47 | 47 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.6 (3.8) | 24.3 (4.3) | 24.5 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 33 | 31 | 64
Region of Enrollment [Number; unit: participants]
  United Kingdom | 47 | 47 | 94

OUTCOME MEASURES:

1. Primary Outcome: Change in LogMAR Corrected Distance Visual Acuity (CDVA)
Description: Change in spectacle corrected logarithm minimum angle of resolution (LogMAR) distance visual acuity recorded in a 4m testing lane in photopic lighting conditions between baseline measurement and final review at 24 months (note that negative change = better vision; 0.1 logMAR units = 1 line on the test chart)
Time Frame: Preoperative vs 24 months
Measure: Mean (Standard Deviation); unit: LogMAR CDVA
Groups:
- CXL Only: CXL only (no PRK) using manual corneal epithelial removal and the same accelerated pulsed protocol as used in the TransPRK group
Arm/Group | TransPRKCXL | CXL Only
Number analyzed (Participants) | 40 | 47
LogMAR CDVA | -0.13 (0.2) | -0.05 (0.13)
Statistical Analysis 1: Comparison: TransPRKCXL vs CXL Only; Null hypothesis = TransPRK produced no gains in vision over and above those produced by CXL only; Test type: Superiority; p = 0.03, t-test, 2 sided

2. Secondary Outcome: Clinically Significant Visual Gain
Description: Number of participants with gain of ≥2 lines (≥0.20 logMAR units) corrected distance visual acuity (CDVA) on a standard 5 letter per line EDTRS visual acuity testing chart
Time Frame: Preoperative vs 24 months postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | TransPRKCXL | CXL Only
Number analyzed (Participants) | 40 | 47
Participants | 12 | 3
Statistical Analysis 1: Comparison: TransPRKCXL vs CXL Only; Null hypothesis = an equal proportion of patients in both study arms have clinically significant visual gains; Test type: Superiority; p = 0.005, Chi-squared

3. Secondary Outcome: Clinically Significant Visual Loss
Description: Number of participants with loss of ≥2 lines (≥0.20 LogMAR units) corrected distance visual acuity (CDVA)
Time Frame: preoperative vs 24 months postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | TransPRKCXL | CXL Only
Number analyzed (Participants) | 40 | 47
Participants | 1 | 2
Statistical Analysis 1: Comparison: TransPRKCXL vs CXL Only; null hypothesis = rates of clinically significant visual loss are equal for TransPRKCXL and CXL only; Test type: Non-Inferiority — Non-inferiority = no significant difference between rates of clinically significant visual loss between groups at the p≤0.05 level; p = 0.13, Chi-squared

4. Secondary Outcome: Change in Kmax - Maximum Local Anterior Corneal Surface Curvature on Tomography Map
Description: Pentacam (www.oculus.de) measure: Maximum local curvature (Kmax). Reduction in dioptric value = corneal flattening
Time Frame: Preoperative vs 24 months postoperative
Measure: Mean (Standard Deviation); unit: Dioptres
Arm/Group | TransPRKCXL | CXL Only
Number analyzed (Participants) | 40 | 47
Dioptres | -5.5 (2.6) | -0.54 (1.6)

5. Secondary Outcome: Progression Rate
Description: The number of participants with possible keratoconus disease progression after treatment defined by a ≥1.5D increase in Kmax, anterior and posterior K2 (maximum local corneal curvature, maximum anterior and posterior meridional corneal curvature) measured using a Pentacam HD corneal tomographer (www.oculus.de).
Time Frame: 6 months postoperative - 24 months postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | TransPRKCXL | CXL Only
Number analyzed (Participants) | 39 | 37
Participants | 3 | 3

ADVERSE EVENTS:
Time Frame: 2 years following the intervention
Groups:
- CXL Only: Standard accelerated corneal collagen cross-linking (historical controls)
  Corneal Collagen Cross-Linking (CXL): Riboflavin soak: 10 minutes total soak time; application of 0.1% riboflavin preparation (VibeX Rapid - www.avedro.com) each 2 minutes with gentle balanced salt solution irrigation to remove excess riboflavin prior to UV light exposure.
  UV light exposure: Total treatment time 8 minutes (370nm wavelength; 30mW/cm2 irradiance; 4 minutes total UV exposure time, pulsed 1.5 seconds on 1.5 seconds off; Avedro KXL I light source)
Arm/Group | TransPRKCXL | CXL Only
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/47
Other Adverse Events (participants affected / at risk) | 1/47 | 0/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TransPRKCXL (N=47) | CXL Only (N=47)
Corneal Infection (Eye disorders) | 1 (1) | 0 (0) — One patient did not attend early follow up and reported to the casualty service 3 weeks after surgery with a bandage contact lens still in situ and corneal infection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes